CLINICAL TRIAL: NCT02653001
Title: Stool Sample Collection for Research Using the In-vitro QIB Colon Model
Brief Title: The QIB Colon Model
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IFR01/2015
Record Dates: First submitted 2016-01-05; First posted 2016-01-12 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Human Gut Microbiota

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): Stool sample collection: Stool samples collected from study participants will be introduced into the colon model to enhance our understanding of the colonic bacterial ecosystem in response to various food components, drugs or biological therapies, and/or to allow investigation the impact of the bacterial ecosystem itself on these added components
  Interventions: Other: Stool sample collection

INTERVENTIONS:
Other: Stool sample collection — Collection of complete stool sample

SUMMARY:
The aim of this project is to establish a list of volunteers willing and able to donate stool samples for use in the model colon so as to facilitate research directed toward understanding the basic science underlying the interactions between the gut microbiome, potential external modifiers, and health.

DETAILED DESCRIPTION:
Adult volunteers will be recruited to donate stool samples for laboratory-based experiments. Once the sample has arrived at QIB 50-100g will be added to the colon model and, depending on the system used, either cultured for 24h or for up to 40 days. During this time, factors under investigation will be added to the model.

Samples added mimic food chyme arriving at the ileal-caecal valve in the intestinal tract. At this stage digested, but non-absorbed food components plus cells and mucous shed from the lining of the small intestine enter the large intestine. Samples of bacteria and media can be taken at any point during the incubation.

Two models are used

1. a simple batch culture in which bacteria, media and test compounds are added to a single compartment and analysed over 24h
2. a three compartment model with continuous flow of media, test compounds and bacteria from the entrance port of the first chamber to the exit of the third chamber mimicking movement through the three main compartments of the colon. This model allows for a stable bacterial population to be established before addition of test compounds, and can remain viable for up to 40 days. In the case of these longer incubations, multiple time points can allow for quite complex experiments looking at interactions between bacteria, food and pharmaceutical products where different factors are added at different time points.

Samples collected during the incubation will be analysed by centrifuging the sample to create a pellet containing bacteria and a supernatant containing a wide range of metabolites. The bacteria will be analysed by extracting their DNA for genomic analysis or using RNA based approaches. On occasion, conventional microbiological techniques might be used. The supernatant will be filter sterilised prior to analysis of its chemical composition by techniques such as mass spectrometry, gel electrophoresis, or chromatography. Alternatively the supernatant may be added to cell lines to model the interaction between the bacterial ecosystem and the cells lining the colon.

ELIGIBILITY:
Inclusion Criteria:

* Live or work within 10 miles of the Norwich Research Park.
* Having a normal bowel habit; assessed as regular defecation between 3 times a day and 3 times a week, with a form similar to 3-5 on the Bristol Stool Chart.
* Do not have any diagnosed chronic gastrointestinal health problem, such as irritable bowel syndrome, inflammatory bowel disease, or coeliac disease.

Exclusion Criteria:

This will depend on individual experiments but in most cases samples will not be collected from individuals:

* who have used antibiotics or probiotics in the last 2 months.
* who are pregnant or breast feeding.
* who have recently used other medications or food supplements (considered on a study-specific basis).
* who have recently had an operation requiring general anaesthetic.
* who have had a gastrointestinal upset, such as vomiting or diarrhoea within the last 72hrs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-12-18 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of 16S rDNA gene (%) | Across an initial period of ten years
  Measurement of 16S rDNA gene in human stool samples will reflect the bacterial population of the colon.

SECONDARY OUTCOMES:
Methane concentration (mmol/L) | Across an initial period of ten years
  Measurement of methane concentration in gaseous production of human stool samples in colon model.
Concentration of short chain fatty acids (mM) | Across an initial period of ten years
  Concentration of short chain fatty acids in the colon model milieu.
Glucosinolate concentration (mM) | Across an initial period of ten years
  Concentration of glucosinolates in the colon model milieu.
Fiber concentration (mM) | Across an initial period of ten years
  Concentration of fiber in the colon model milieu.

CONTACTS AND LOCATIONS:
Overall Officials: Arjan Narbad, Ph.D, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Quadram Institute Bioscience, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Day-Walsh P, Shehata E, Saha S, Savva GM, Nemeckova B, Speranza J, Kellingray L, Narbad A, Kroon PA. The use of an in-vitro batch fermentation (human colon) model for investigating mechanisms of TMA production from choline, L-carnitine and related precursors by the human gut microbiota. Eur J Nutr. 2021 Oct;60(7):3987-3999. doi: 10.1007/s00394-021-02572-6. Epub 2021 May 2. PMID 33934200